CLINICAL TRIAL: NCT03130855
Title: Buccal Infiltration Technique Compared to Inferior Alveolar Nerve Block Technique for Alleviation of Intraoperative Pain During Pulpal Treatment of Mandibular Primary Molars: A Randomized Controlled Clinical Trial.
Brief Title: Comparison Between Efficiency of Inferior Alveolar Nerve Block and Buccal Infiltration Techniques Using Articaine 4% 1:100000
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Sherif Ahmed Abo El Abbas, resident at pediatric dentistry and public health faculty of oral and dental medicine cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: articaine
Record Dates: First submitted 2017-04-02; First posted 2017-04-27 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Anesthesia, Local
Keywords: pediatric patients; articaine local anesthesia
MeSH Terms: interventions — Carticaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inferior alveolar nerve block with 4% articaine (Experimental): inferior alveolar nerve block using 4% articaine anesthetic solution
  Interventions: Drug: inferior alveolar nerve block with 4% articaine
- buccal infiltration with 4% articaine (Active Comparator): buccal infiltration using 4% articaine anesthetic solution
  Interventions: Drug: buccal infiltration with 4% articaine

INTERVENTIONS:
Drug: inferior alveolar nerve block with 4% articaine — an anesthetic technique using 4% articaine anesthetic solution
  Arms: inferior alveolar nerve block with 4% articaine
Drug: buccal infiltration with 4% articaine — anesthetic technique using 4% articaine anesthetic solution
  Arms: buccal infiltration with 4% articaine

SUMMARY:
This split mouth randomized control trial is designed as to compare the effectiveness of the buccal infiltration technique with the gold standard inferior alveolar nerve block in anesthetizing mandibular second primary molars to undergoing pulpal treatment.

patient will be videotaped during pulpal treatment of their teeth and an accessing pain will be through an objective pain scale (SEM scale), (sound-eye-motor scale).

the patient will be asked to fill in a subjective Wong Baker pain scale for the pain suffered during injecting the local anesthetic agent in both techniques.

ELIGIBILITY:
A-Inclusion Criteria:

1. first dental visit.
2. cooperative children (rating 4 or 3 based on Frankl behavior scale) aging from 6 to 8 years suffering from one or more deep carious lesions in their primary molars seeking treatment.
3. Restorable molars with stainless steel crowns.

B-Exclusion Criteria:

1. medically compromised patients. uncooperative children (rating 1 or 2 on the Frankl behavior scale)needing special line of treatment through general anesthesia.
2. signs and symptoms of irreversible pulpitis, spontaneous pain, necrosis or any signs or symptoms of any infection.
3. presence of any radiographic signs of abcess, bone loss, internal or external root resorption.
4. parents or guardians who refuse participating in the study.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2017-05-15 (Estimated); Primary Completion 2017-07-01 (Estimated); Study Completion 2017-08-01 (Estimated)

PRIMARY OUTCOMES:
pain experienced by child during pulpal treatment | one week
  sound-eye-motor

SECONDARY OUTCOMES:
time needed for numbness | one week
  stop watch
pain experienced by the child due to needle prick | one week
  Wong Baker facial pain scale

IPD SHARING:
Plan to Share IPD: No